CLINICAL TRIAL: NCT00145522
Title: A Twelve 28-Day Cycles, Multicenter, Prospective, Randomized, Open, Blinded Endpoint, Parallel Group Study Comparing the Effect on Breast and Cardiovascular Metabolic Markers of Continuously Combined 17β-Estradiol/Dydrogesterone and Tibolone in Postmenopausal Women.
Brief Title: Study to Compare the Effect of Hormone Replacement Therapy (HRT) on Breast and Cardiovascular Metabolic Markers in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: Irene Grazioli, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S102.4.103; 2004-001829-22
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Menopause
Keywords: Menopause, IGF-1, HRT
MeSH Terms: interventions — Dydrogesterone; tibolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: 17ß-Estradiol/Dydrogesterone
- 2 (Active Comparator)
  Interventions: Drug: Tibolone

INTERVENTIONS:
Drug: 17ß-Estradiol/Dydrogesterone — 1/5 mg/day for 12 cycles of 28 days
  Arms: 1
Drug: Tibolone — 2,5 mg/day for 12 cycles of 28 days
  Arms: 2

SUMMARY:
This study is to evaluate the effects of continuously combined 17b-estradiol/dydrogesterone in comparison with tibolone on the breast metabolic markers, in particular the total insulin-like growth factor-1 (IGF-1), in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Natural or surgical postmenopausal amenorrhea since ≥ 12 months,
* non hysterectomized women, complaining of at least 14 hot flushes per week

Exclusion Criteria:

* Known, suspected or history of breast cancer or hormone-dependent neoplasia,
* undiagnosed genital bleeding,
* venous or arterial history or presence of thromboembolism,
* cerebrovascular disease

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
IGF1 values after 12 cycles of 28 days | 1 year

SECONDARY OUTCOMES:
after 12 cycles of 28 days: other breast metabolic markers [IGFBP 1 and 3, SHBG, free estradiol, fasting insulin], breast tenderness and breast density, cardiovascular metabolic markers, menopausal symptoms and bleeding pattern | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (11):
- Italy (11):
  - Site 8, Ancona
  - Site 15, Cagliari
  - Site 4, Catania
  - Site 9, Florence
  - Site 10, Milan
  - Site 11, Milan
  - Sit 14, Modena
  - Site 6, Roma
  - Site 1, Torino
  - Site 2, Torino
  - Site 7, Udine